CLINICAL TRIAL: NCT06355076
Title: Comparison of New Reconstruction and Anastomosis in Robot-assisted Laparoscopic Radical Resection: a Prospective Randomized Controlled Study
Brief Title: New Urethral Reconstruction in Robot-assisted Laparoscopic Radical Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSZ03
Record Dates: First submitted 2024-03-31; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The experimental group received a new urethral reconstruction technique, which involves suturing the levator ani muscle with the lateral striated muscle of the urethra, the dorsal median ridge (MDR), and the Di's fascia together for continuous suturing before performing bladder urethral anastomosis. After the reconstruction is completed, the end to end anastomosis of the bladder urethra is performed
Who Masked: Participant
Masking Description: Patients in the experimental or control group, as well as their family members, are unaware
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- New urethral reconstruction arm (Experimental): The experimental group received a new reconstruction technique, in which the levator anus and the dorsal median ridge (MDR) of the lateral striated muscle were sutured to the Dirichlet fascia for continuous suture before anastomosis
  Interventions: Procedure: New urethral reconstruction
- Traditional bladder urethral anastomosis arm (Active Comparator): End to end anastomosis of bladder and urethra
  Interventions: Procedure: New urethral reconstruction

INTERVENTIONS:
Procedure: New urethral reconstruction — This kind of reconstruction suture has larger area, higher firmness, better fixation of the position of broken end and prolongation of functional length.

SUMMARY:
The purpose of this clinical trial is to compare new reconstruction and anastomosis in robot-assisted radical laparoscopic resection It will also understand the possibility of exploring new reconstruction in completely solving patients' postoperative urinary incontinence The main questions it aims to answer are:

Is there a significant improvement in urinary control in patients with new reconstruction compared with patients with anastomosis? The researchers compared the new reconstruction with anastomosis in robot-assisted laparoscopic radical resection to see if the new reconstruction improved urinary incontinence after operation.

Participants will:

The intervention group adopted the new reconstruction proposed by our team; End-to-end anastomosis was performed in non-intervention group.

DETAILED DESCRIPTION:
It is one of the most common malignant tumors in urology, and its incidence rate is the second among male malignant tumors in the world. In recent years, with the economic and social development in China, the incidence rate has increased year by year, which seriously threatens the Radical resection is the current treatment plan. Although radical surgery can prolong the survival time of patients, because of the surgical injury, the incidence of urinary incontinence and sexual function after operation is high, which greatly affects the physiological health, mental health and social function of patients.

In order to solve the above problems, Professor Shi Benkang's team of Urology Department of Qilu Hospital of Shandong University improved the existing urinary tract reconstruction after consulting a large number of related literatures and combining with the new findings of our team's previous anatomical work, which needed to be carried out under Da Vinci Xi surgical system. By continuously suturing the fascia on the surface of levator anal muscle and the posterior dorsal median ridge (MDR) and Dirichlet fascia of the lateral tissue, it achieved the purpose of protecting the apical saccular tube bundle (NVB) and maintaining the stability of the length of vascular and nerve lengthening function in the posterior MDR We found that the postoperative urinary incontinence of patients with new reconstruction technique is obviously better than that of anastomosis, which provides a new idea for improving the postoperative urinary incontinence of RARP patients.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years old, confirmed by puncture pathology as prostate cancer
* The tumor has no extensive distant metastasis, or has reached a resectable state through neoadjuvant chemotherapy and endocrine therapy
* Willing to accept robot assisted laparoscopic radical prostatectomy

Exclusion criteria:

* Tumor metastasis cannot achieve curative effect through surgery
* Concomitant severe cardiovascular and cerebrovascular complications
* Merge severe mental and neurological disorders
* Poor liver and kidney function
* Refusal to accept robot assisted laparoscopic radical prostatectomy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-02-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Recovery of urinary incontinence | at the first time of catheter extubation, 1 month, 3 months, 6 months and 1 year after catheter extubation
  Recovery of urinary incontinence in intervention group and non-intervention group at the first time of catheter extubation, 1 month, 3 months, 6 months and 1 year after catheter extubation

SECONDARY OUTCOMES:
complication | at the first time of catheter extubation, 1 month, 3 months, 6 months and 1 year after catheter extubation
  complications include infection, bleeding, etc.
PSA | at the first time of catheter extubation, 1 month, 3 months, 6 months and 1 year after catheter extubation
  Prostate Specific Antigen
recurrence | at the first time of catheter extubation, 1 month, 3 months, 6 months and 1 year after catheter extubation
  Tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Shouzhen Chen, Dr., Study Chair — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital, Jinan, Shandong, China

REFERENCES:
- [Background] Ficarra V, Rossanese M, Crestani A, Alario G, Mucciardi G, Isgro A, Giannarini G. Robot-assisted Radical Prostatectomy Using the Novel Urethral Fixation Technique Versus Standard Vesicourethral Anastomosis. Eur Urol. 2021 Apr;79(4):530-536. doi: 10.1016/j.eururo.2021.01.028. Epub 2021 Feb 4. PMID 33551295
- [Background] Cui J, Guo H, Li Y, Chen S, Zhu Y, Wang S, Wang Y, Liu X, Wang W, Han J, Chen P, Nie S, Yin G, Shi B. Pelvic Floor Reconstruction After Radical Prostatectomy: A Systematic Review and Meta-analysis of Different Surgical Techniques. Sci Rep. 2017 Jun 2;7(1):2737. doi: 10.1038/s41598-017-02991-8. PMID 28578433
- [Background] Rocco B, Gregori A, Stener S, Santoro L, Bozzola A, Galli S, Knez R, Scieri F, Scaburri A, Gaboardi F. Posterior reconstruction of the rhabdosphincter allows a rapid recovery of continence after transperitoneal videolaparoscopic radical prostatectomy. Eur Urol. 2007 Apr;51(4):996-1003. doi: 10.1016/j.eururo.2006.10.014. Epub 2006 Oct 23. PMID 17079070
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103
- [Background] Mungovan SF, Carlsson SV, Gass GC, Graham PL, Sandhu JS, Akin O, Scardino PT, Eastham JA, Patel MI. Preoperative exercise interventions to optimize continence outcomes following radical prostatectomy. Nat Rev Urol. 2021 May;18(5):259-281. doi: 10.1038/s41585-021-00445-5. Epub 2021 Apr 8. PMID 33833445
- [Result] Moore K, Allen M, Voaklander DC. Pad tests and self-reports of continence in men awaiting radical prostatectomy: establishing baseline norms for males. Neurourol Urodyn. 2004;23(7):623-6. doi: 10.1002/nau.20067. PMID 15382185
- [Result] Qi W, Dou M, Xu L, Qu S, Zhu Y, Chen S, Shi B. Robot-assisted radical prostatectomy using a novel urethral reconstruction technique vs standard vesicourethral anastomosis. A retrospective cohort study. World J Urol. 2023 Jan;41(1):51-58. doi: 10.1007/s00345-022-04208-8. Epub 2022 Nov 24. PMID 36434138